CLINICAL TRIAL: NCT00434577
Title: A Phase II, Single-blind, Randomized, Controlled, Multicentre Vaccination Study to Evaluate the Safety and Immune Response of the GSK Biologicals Zoster Vaccine, gE/AS01B, and to Compare 3 Doses of gE With AS01B Adjuvant in Healthy Elderly Subjects, Aged 60 to 69 Years and 70 Years and Above.
Brief Title: Safety and Immunogenicity of the Zoster Vaccine GSK1437173A in Elderly Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 108494; 108516 (Other: GSK); 108518 (Other: GSK); 108520 (Other: GSK); 2006-004863-69 (EudraCT Number)
Record Dates: First submitted 2007-02-12; First posted 2007-02-13 (Estimated); Results first posted 2019-01-08 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-02

CONDITIONS: Herpes Zoster
Keywords: GSK Biologicals; Herpes Zoster (HZ); Vaccine; Varicella Zoster Virus (VZV); Shingles
MeSH Terms: conditions — Herpes Zoster; Chickenpox

STUDY DESIGN:
Who Masked: Participant

ARMS (5):
- GSK1437173A _LD Group (Experimental): Healthy male or female subjects aged 60 years or older, who received 2 doses of herpes zoster subunit vaccine (GSK1437173A) low dose (LD) formulation, according to a 0, 2-month schedule. The vaccine was administrated by intramuscular injection (IM) in the upper deltoid site of the left arm.
  Interventions: Biological: Herpes Zoster vaccine GSK1437173A Low Dose
- GSK1437173A _MD Group (Experimental): Healthy male or female subjects aged 60 years or older, who received 2 doses of herpes zoster subunit vaccine (GSK1437173A) medium dose (MD) formulation, according to a 0, 2-month schedule. The vaccine was administrated by (IM) in the upper deltoid site of the left arm.
  Interventions: Biological: Herpes Zoster vaccine GSK1437173A Medium Dose
- GSK1437173A _HD Group (Experimental): Healthy male or female subjects aged 60 years or older, who received 2 doses of herpes zoster subunit vaccine (GSK1437173A) high dose (HD) formulation, according to a 0, 2-month schedule. The vaccine was administrated by (IM) in the upper deltoid site of the left arm.
  Interventions: Biological: Herpes Zoster vaccine GSK1437173A High Dose
- Placebo + GSK1437173A _HD Group (Placebo Comparator): Healthy male or female subjects aged 60 years or older, who received a 1st dose of saline solution and a 2nd dose of GSK1437173A high dose (HD) formulation, according to a 0, 2-month schedule. The vaccine was administrated by (IM) in the upper deltoid site of the left arm.
  Interventions: Biological: Herpes Zoster vaccine GSK1437173A High Dose; Biological: Placebo
- GSK1437173A_MODIFIED GROUP (Active Comparator): Healthy male or female subjects aged 60 years or older, who received 2 doses of GSK1437173A modified formulation vaccine reconstituted with saline solution, according to a 0, 2-month schedule. The vaccine was administrated by (IM) in the upper deltoid site of the left arm.
  Interventions: Biological: Herpes Zoster vaccine GSK1437173A Modified

INTERVENTIONS:
Biological: Herpes Zoster vaccine GSK1437173A Low Dose — Single or two-dose intramuscular injection.
  Arms: GSK1437173A _LD Group
Biological: Herpes Zoster vaccine GSK1437173A Medium Dose — Single or two-dose intramuscular injection.
  Arms: GSK1437173A _MD Group
Biological: Herpes Zoster vaccine GSK1437173A High Dose — Single or two-dose intramuscular injection.
  Arms: GSK1437173A _HD Group; Placebo + GSK1437173A _HD Group
Biological: Herpes Zoster vaccine GSK1437173A Modified — Single or two-dose intramuscular injection.
  Arms: GSK1437173A_MODIFIED GROUP
Biological: Placebo — Single intramuscular injection
  Arms: Placebo + GSK1437173A _HD Group

SUMMARY:
Based on the results of a previous clinical PhaseI/II study, GSK1437173A is the lead GSK candidate Herpes Zoster (HZ) vaccine to prevent episodes of HZ (shingles). This phase II study will be subdivided into a primary study (108494) and three extension studies (108516, 108518 & 108520), consisting of one additional visit each at months 12, 24 and 36, respectively, from the first visit of the Zoster-003 primary study onwards. The aim of the primary 108494 study is to evaluate the immunogenicity & safety of different dosages of the GSK1437173A vaccine in healthy elderly population. The study population will be stratified by age. The primary objective of this trial is to select the best dosage of GSK1437173A. The aim of the extension studies is to evaluate the persistence of the immune response induced by the candidate HZ vaccine during a long term period.

No new subjects will be enrolled during the extension phases of the study.

DETAILED DESCRIPTION:
The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol.
* A male or female aged 60 years or older at the time of the first vaccination.
* Written informed consent obtained from the subject

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first injection with study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs during the study period, except inhaled and topical steroids are allowed.
* Administration or planned administration of a vaccine not foreseen by the study protocol within 2 weeks of the first study vaccine injection, with the exception of the influenza vaccine, which can be administered 1 week preceding or 1 month after the first study vaccine injection.
* Previous vaccination against HZ.
* History of herpes zoster (Shingles).
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Acute disease at the time of enrolment.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by subject's medical history or physical examination as assessed by the investigator.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the first injection of study vaccine or planned administration during the study period.
* History of or current drug and/or alcohol abuse.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 715 (Actual)
Dates: Start 2007-02-14 (Actual); Primary Completion 2007-10-04 (Actual); Study Completion 2010-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (11):
- GSK Investigational Site, Hradec Králové, Czechia
- Germany (6):
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Berlin
- Netherlands (2):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Rotterdam
- Sweden (2):
  - GSK Investigational Site, Eskilstuna
  - GSK Investigational Site, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Chlibek R, Smetana J, Pauksens K, Rombo L, Van den Hoek JA, Richardus JH, Plassmann G, Schwarz TF, Ledent E, Heineman TC. Safety and immunogenicity of three different formulations of an adjuvanted varicella-zoster virus subunit candidate vaccine in older adults: a phase II, randomized, controlled study. Vaccine. 2014 Mar 26;32(15):1745-53. doi: 10.1016/j.vaccine.2014.01.019. Epub 2014 Feb 6. PMID 24508036
- [Derived] Schwarz TF, Volpe S, Catteau G, Chlibek R, David MP, Richardus JH, Lal H, Oostvogels L, Pauksens K, Ravault S, Rombo L, Sonder G, Smetana J, Heineman T, Bastidas A. Persistence of immune response to an adjuvanted varicella-zoster virus subunit vaccine for up to year nine in older adults. Hum Vaccin Immunother. 2018 Jun 3;14(6):1370-1377. doi: 10.1080/21645515.2018.1442162. Epub 2018 Mar 21. PMID 29461919
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 108494 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 108494 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 108494 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 108494 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 108494 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 108494 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 108494 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 715 subjects enrolled, only 714 were vaccinated.
Period: Months 0-3
Arm/Group | GSK1437173A _LD Group | GSK1437173A _MD Group | GSK1437173A _HD Group | Placebo + GSK1437173A _HD Group | GSK1437173A_MODIFIED Group
Started | 164 | 166 | 165 | 165 | 54
Completed | 161 | 164 | 161 | 164 | 51
Not Completed | 3 | 2 | 4 | 1 | 3
Not completed — Serious Adverse Event | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 2
Not completed — Protocol Violation | 1 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 1 | 1
Period: Month 12
Arm/Group | GSK1437173A _LD Group | GSK1437173A _MD Group | GSK1437173A _HD Group | Placebo + GSK1437173A _HD Group | GSK1437173A_MODIFIED Group
Started | 156 | 159 | 159 | 161 | 50
Completed | 156 | 159 | 159 | 161 | 50
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Month 24
Arm/Group | GSK1437173A _LD Group | GSK1437173A _MD Group | GSK1437173A _HD Group | Placebo + GSK1437173A _HD Group | GSK1437173A_MODIFIED Group
Started | 150 | 155 | 154 | 157 | 49
Completed | 150 | 155 | 154 | 157 | 49
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Month 36
Arm/Group | GSK1437173A _LD Group | GSK1437173A _MD Group | GSK1437173A _HD Group | Placebo + GSK1437173A _HD Group | GSK1437173A_MODIFIED Group
Started | 147 | 147 | 150 | 155 | 47
Completed | 147 | 147 | 150 | 155 | 47
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK1437173A _LD Group | GSK1437173A _MD Group | GSK1437173A _HD Group | Placebo + GSK1437173A _HD Group | GSK1437173A_MODIFIED GROUP | Total
Number analyzed (Participants) | 164 | 166 | 165 | 165 | 54 | 714
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.8 (5.5) | 72.9 (5.1) | 73.0 (5.7) | 73.1 (5.9) | 72.1 (5.2) | 72.9 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 100 | 85 | 95 | 36 | 404
  Male | 76 | 66 | 80 | 70 | 18 | 310
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Geographic ancestry: African Heritage/African American | 0 | 1 | 0 | 0 | 0 | 1
  Geographic ancestry: Asian - Central/South Asian Heritage | 0 | 1 | 0 | 0 | 0 | 1
  Geographic ancestry: White - Arabic/North African Heritage | 1 | 1 | 1 | 0 | 0 | 3
  Geographic ancestry: White - Caucasian/European Heritage | 162 | 163 | 164 | 165 | 54 | 708
  Geographic ancestry: Other | 1 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Glycoprotein E (gE)-Specific Cluster of Differentiation (CD4) T-cells Expressing at Least Two Different Activation Markers
Description: Among the activation markers expressed were interleukin-2 [IL-2] and/or interferon-gamma [IFN-γ] and/or tumour necrosis factor-alpha [TNF-α] and/or cluster of differentiation 40-ligand [CD40-L]. Analysis of cytokines expression was done by means of in vitro flow cytometry using intracellular cytokine staining (ICS) in subjects aged 70 or higher (≥).
Time Frame: One month after the second vaccination (Month 3)
Population: The analysis was performed on the According-to-Protocol(ATP) cohort for Immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available.
Measure: Median (Inter-Quartile Range); unit: T-cells/million cells
Arm/Group | GSK1437173A _LD Group | GSK1437173A _MD Group | GSK1437173A _HD Group | Placebo + GSK1437173A _HD Group | GSK1437173A_MODIFIED Group
Number analyzed (Participants) | 119 | 120 | 117 | 118 | 36
T-cells/million cells | 1801.23 [907.17 to 2930.71] | 1722.83 [1172.96 to 3229.73] | 1778.48 [1154.88 to 3407.91] | 491.03 [320.65 to 768.17] | 388.49 [208.57 to 610.66]

2. Primary Outcome: Frequency Odds Ratio of gE-specific CD4 T-cells Expressing at Least Two Different Activation Markers
Description: Among the activation markers expressed were interleukin-2 [IL-2] and/or interferon-gamma [IFN-γ] and/or tumour necrosis factor-alpha [TNF-α] and/or cluster of differentiation 40-ligand [CD40-L]. Analysis of cytokines expression was done by means of in vitro flow cytometry using intracellular cytokine staining (ICS) in subjects ≥ 70 years old. The odds-ratios are calculated using the the frequency of CD4 secreting cytokines, upon in vitro stimulation with the specific antigen, at the numerator and the frequency of the CD4 secreting cytokines with the medium only (background level) at the denominator. The odds-ratios represent the fold-change in the specific response compared to the background level.
Time Frame: One month after the second vaccination (Month 3)
Population: The analysis was performed on the ATP cohort for Immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available.
Measure: Mean (Standard Deviation); unit: Fold Change
Arm/Group | GSK1437173A _LD Group | GSK1437173A _MD Group | GSK1437173A _HD Group | Placebo + GSK1437173A _HD Group | GSK1437173A_MODIFIED Group
Number analyzed (Participants) | 119 | 120 | 117 | 118 | 36
Fold Change | 12.83 (13.13) | 15.00 (15.86) | 21.53 (71.96) | 5.92 (9.56) | 4.05 (3.20)

3. Primary Outcome: Frequency of gE-specific CD4 T-cells Expressing at Least Two Different Activation Markers
Description: Among the activation markers expressed were interleukin-2 [IL-2] and/or interferon-gamma [IFN-γ] and/or tumour necrosis factor-alpha [TNF-α] and/or cluster of differentiation 40-ligand [CD40-L]. Analysis of cytokines expression was done by means of in vitro flow cytometry using intracellular cytokine staining (ICS) in subjects ≥ 70 years old.
Time Frame: One month after the second vaccination (Month 3)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-cells/million cells
Arm/Group | GSK1437173A _LD Group | GSK1437173A _MD Group | GSK1437173A _HD Group | Placebo + GSK1437173A _HD Group | GSK1437173A_MODIFIED Group
Number analyzed (Participants) | 119 | 120 | 117 | 118 | 36
T-cells/million cells | 2269.84 (1934.55) | 2441.95 (2055.11) | 2449.90 (1808.00) | 681.73 (665.17) | 512.55 (463.35)

4. Secondary Outcome: Frequency of gE-specific CD4 T-cells Expressing at Least Two Different Activation Markers
Description: Among the activation markers expressed were interleukin-2 [IL-2] and/or interferon-gamma [IFN-γ] and/or tumour necrosis factor-alpha [TNF-α] and/or cluster of differentiation 40-ligand [CD40-L]. Analysis of cytokines expression was done by means of in vitro flow cytometry using intracellular cytokine staining (ICS) in subjects 60 to 69 years (60-69y) and ≥ 70 years (+70y) old.
Time Frame: At pre-vaccination (Day 0), one month after the first vaccination (Month 2) and second vaccination (Month 3)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-cells/million cells
Arm/Group | GSK1437173A _LD Group | GSK1437173A _MD Group | GSK1437173A _HD Group | Placebo + GSK1437173A _HD Group | GSK1437173A_MODIFIED Group
Number analyzed (Participants) | 152 | 150 | 144 | 150 | 48
T-cells/million cells
  CD4-All Doubles, Day 0: number analyzed (Participants) | 152 | 146 | 142 | 149 | 48
  CD4-All Doubles, Day 0 | 194.47 (214.96) | 225.47 (370.67) | 201.17 (230.96) | 203.70 (221.97) | 145.95 (164.57)
  CD4-All Doubles, Month 2: number analyzed (Participants) | 152 | 150 | 142 | 150 | 48
  CD4-All Doubles, Month 2 | 459.01 (401.25) | 482.84 (425.73) | 489.45 (423.52) | 173.91 (181.86) | 230.28 (250.70)
  CD4-All Double, Month 3: number analyzed (Participants) | 151 | 148 | 144 | 148 | 47
  CD4-All Double, Month 3 | 2246.29 (1976.42) | 2372.07 (1877.43) | 2569.29 (2052.74) | 670.80 (606.93) | 550.11 (448.15)

5. Secondary Outcome: Frequency of gE-specific CD4 T-cells Expressing IFN-γ and at Least Another Activation Marker
Description: Among other activation markers expressed were interleukin-2 [IL-2] or tumour necrosis factor-alpha [TNF-α] or cluster of differentiation 40-ligand [CD40-L]. Analysis of cytokines expression was done by means of in vitro flow cytometry using intracellular cytokine staining (ICS).
Time Frame: At pre-vaccination (Day 0), one month after the first vaccination (Month 2) and second vaccination (Month 3)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-cells/million cells
Arm/Group | GSK1437173A _LD Group | GSK1437173A _MD Group | GSK1437173A _HD Group | Placebo + GSK1437173A _HD Group | GSK1437173A_MODIFIED Group
Number analyzed (Participants) | 151 | 150 | 144 | 148 | 48
T-cells/million cells
  Day 0: number analyzed (Participants) | 149 | 144 | 139 | 148 | 48
  Day 0 | 156.54 (199.12) | 169.01 (326.34) | 152.28 (220.50) | 157.13 (180.00) | 118.35 (125.08)
  Month 2: number analyzed (Participants) | 151 | 150 | 142 | 147 | 46
  Month 2 | 279.39 (343.61) | 279.20 (336.29) | 292.15 (345.65) | 124.05 (151.42) | 168.34 (213.83)
  Month 3: number analyzed (Participants) | 151 | 148 | 144 | 148 | 46
  Month 3 | 1179.29 (1021.14) | 1296.04 (1132.18) | 1417.40 (1303.60) | 363.23 (364.74) | 341.36 (313.79)

6. Secondary Outcome: Frequency of gE-specific CD4 T-cells Expressing IL-2 and at Least Another Activation Marker
Description: Among other activation markers expressed were interferon-gamma [IFN-γ] or tumour necrosis factor-alpha [TNF-α] or cluster of differentiation 40-ligand [CD40-L]. Analysis of cytokines expression was done by means of in vitro flow cytometry using intracellular cytokine staining (ICS).
Time Frame: At pre-vaccination (Day 0), one month after the first vaccination (Month 2) and second vaccination (Month 3)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-cells/million cells
Arm/Group | GSK1437173A _LD Group | GSK1437173A _MD Group | GSK1437173A _HD Group | Placebo + GSK1437173A _HD Group | GSK1437173A_MODIFIED Group
Number analyzed (Participants) | 152 | 150 | 144 | 150 | 48
T-cells/million cells
  Day 0: number analyzed (Participants) | 152 | 146 | 142 | 149 | 48
  Day 0 | 171.21 (208.49) | 191.28 (307.40) | 180.85 (193.48) | 172.41 (184.32) | 125.22 (134.81)
  Month 2: number analyzed (Participants) | 152 | 150 | 142 | 150 | 48
  Month 2 | 416.12 (369.85) | 442.17 (363.10) | 438.27 (378.81) | 150.47 (160.29) | 199.34 (224.39)
  Month 3: number analyzed (Participants) | 151 | 148 | 144 | 148 | 47
  Month 3 | 2077.06 (1860.40) | 2156.40 (1697.78) | 2315.84 (1847.24) | 597.76 (531.07) | 491.06 (396.39)

7. Secondary Outcome: Frequency of gE-specific CD4 T-cells Expressing TNF-α and at Least Another Activation Marker
Description: Among other activation markers expressed were interleukin-2 [IL-2] or interferon-gamma [IFN-γ] or cluster of differentiation 40-ligand [CD40-L]. Analysis of cytokines expression was done by means of in vitro flow cytometry using intracellular cytokine staining (ICS).
Time Frame: At pre-vaccination (Day 0), one month after the first vaccination (Month 2) and second vaccination (Month 3)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-cells//million cells
Arm/Group | GSK1437173A _LD Group | GSK1437173A _MD Group | GSK1437173A _HD Group | Placebo + GSK1437173A _HD Group | GSK1437173A_MODIFIED Group
Number analyzed (Participants) | 152 | 150 | 144 | 150 | 48
T-cells//million cells
  Day 0: number analyzed (Participants) | 152 | 144 | 141 | 149 | 48
  Day 0 | 97.28 (137.06) | 121.05 (296.79) | 116.91 (173.65) | 110.66 (162.02) | 81.40 (107.44)
  Month 2: number analyzed (Participants) | 152 | 150 | 142 | 150 | 47
  Month 2 | 251.94 (277.71) | 256.15 (304.91) | 263.39 (284.96) | 95.84 (125.15) | 120.73 (148.24)
  Month 3: number analyzed (Participants) | 151 | 148 | 144 | 148 | 47
  Month 3 | 1317.39 (1304.53) | 1282.96 (1183.69) | 1389.62 (1231.76) | 350.23 (380.60) | 252.86 (253.55)

8. Secondary Outcome: Frequency of gE-specific CD4 T-cells Expressing CD40L and at Least Another Activation Marker
Description: Among other activation markers expressed were interleukin-2 [IL-2] or interferon-gamma [IFN-γ] or tumour necrosis factor-alpha [TNF-α] . Analysis of cytokines expression was done by means of in vitro flow cytometry using intracellular cytokine staining (ICS).
Time Frame: At pre-vaccination (Day 0), one month after the first vaccination (Month 2) and second vaccination (Month 3)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-cells/million cells
Arm/Group | GSK1437173A _LD Group | GSK1437173A _MD Group | GSK1437173A _HD Group | Placebo + GSK1437173A _HD Group | GSK1437173A_MODIFIED Group
Number analyzed (Participants) | 152 | 150 | 144 | 149 | 48
T-cells/million cells
  Day 0: number analyzed (Participants) | 152 | 144 | 142 | 149 | 48
  Day 0 | 142.88 (169.52) | 153.80 (214.95) | 151.37 (160.38) | 155.90 (187.47) | 111.55 (126.92)
  Month 2: number analyzed (Participants) | 152 | 150 | 142 | 149 | 48
  Month 2 | 385.34 (348.25) | 405.95 (359.46) | 417.20 (361.59) | 132.62 (144.06) | 182.82 (195.36)
  Month 3: number analyzed (Participants) | 151 | 148 | 144 | 148 | 47
  Month 3 | 2014.37 (1849.25) | 2154.81 (1799.64) | 2303.13 (1987.94) | 567.33 (566.48) | 433.56 (391.64)

9. Secondary Outcome: Frequency of gE-specific CD8 T-cells Expressing at Least Two Different Activation Markers
Description: Among the activation markers expressed were interleukin-2 [IL-2] and/or interferon-gamma [IFN-γ] and/or tumour necrosis factor-alpha [TNF-α] and/or cluster of differentiation 40-ligand [CD40-L]. Analysis of cytokines expression was done by means of in vitro flow cytometry using intracellular cytokine staining (ICS).
Time Frame: At pre-vaccination (Day 0), one month after the first vaccination (Month 2) and second vaccination (Month 3)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-cells/million cells
Arm/Group | GSK1437173A _LD Group | GSK1437173A _MD Group | GSK1437173A _HD Group | Placebo + GSK1437173A _HD Group | GSK1437173A_MODIFIED Group
Number analyzed (Participants) | 126 | 120 | 118 | 119 | 39
T-cells/million cells
  CD8-All Doubles, Day 0: number analyzed (Participants) | 112 | 117 | 118 | 109 | 32
  CD8-All Doubles, Day 0 | 74.62 (118.02) | 98.88 (164.52) | 122.37 (221.20) | 80.54 (121.84) | 108.21 (330.11)
  CD8-All Doubles, Month 2: number analyzed (Participants) | 102 | 120 | 118 | 108 | 39
  CD8-All Doubles, Month 2 | 85.29 (139.32) | 106.23 (141.63) | 86.35 (168.10) | 120.06 (221.20) | 98.97 (299.34)
  CD8-All Doubles, Month 3: number analyzed (Participants) | 126 | 118 | 112 | 119 | 38
  CD8-All Doubles, Month 3 | 96.43 (155.37) | 88.77 (140.95) | 117.70 (196.09) | 112.99 (165.52) | 116.41 (450.85)

10. Secondary Outcome: Frequency of gE-specific CD8 T-cells Expressing IFN-γ and at Least Another Activation Marker
Description: as for outcome 5
Time Frame: At pre-vaccination (Day 0), one month after the first vaccination (Month 2) and second vaccination (Month 3)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-cells/million cells
Arm/Group | GSK1437173A _LD Group | GSK1437173A _MD Group | GSK1437173A _HD Group | Placebo + GSK1437173A _HD Group | GSK1437173A_MODIFIED Group
Number analyzed (Participants) | 98 | 91 | 98 | 95 | 32
T-cells/million cells
  Day 0: number analyzed (Participants) | 94 | 90 | 95 | 92 | 26
  Day 0 | 60.35 (97.12) | 75.79 (114.55) | 106.39 (199.96) | 70.69 (121.23) | 123.99 (360.75)
  Month 2: number analyzed (Participants) | 87 | 87 | 98 | 90 | 30
  Month 2 | 65.97 (111.02) | 106.74 (133.15) | 72.58 (92.99) | 106.02 (184.40) | 95.05 (326.45)
  Month 3: number analyzed (Participants) | 98 | 91 | 97 | 95 | 32
  Month 3 | 88.62 (136.13) | 76.92 (123.74) | 95.01 (138.77) | 96.91 (161.10) | 125.69 (480.05)

11. Secondary Outcome: Frequency of gE-specific CD8 T-cells Expressing IL-2 and at Least Another Activation Marker
Description: as for outcome 6
Time Frame: At pre-vaccination (Day 0), one month after the first vaccination (Month 2) and second vaccination (Month 3)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-cells/million cells
Arm/Group | GSK1437173A _LD Group | GSK1437173A _MD Group | GSK1437173A _HD Group | Placebo + GSK1437173A _HD Group | GSK1437173A_MODIFIED Group
Number analyzed (Participants) | 97 | 91 | 88 | 90 | 27
T-cells/million cells
  Day 0: number analyzed (Participants) | 74 | 79 | 84 | 78 | 27
  Day 0 | 81.42 (108.62) | 83.13 (131.07) | 90.71 (140.18) | 63.56 (89.18) | 43.03 (58.88)
  Month 2: number analyzed (Participants) | 72 | 86 | 78 | 81 | 25
  Month 2 | 61.05 (106.36) | 78.18 (92.65) | 83.07 (186.88) | 82.47 (126.08) | 68.98 (85.29)
  Month 3: number analyzed (Participants) | 97 | 91 | 88 | 90 | 26
  Month 3 | 69.06 (97.12) | 65.08 (83.71) | 103.17 (179.57) | 82.95 (99.47) | 56.42 (120.85)

12. Secondary Outcome: Frequency of gE-specific CD8 T-cells Expressing TNF-α and at Least Another Activation Marker
Description: as for outcome 7
Time Frame: At pre-vaccination (Day 0), one month after the first vaccination (Month 2) and second vaccination (Month 3)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-cells/million cells
Arm/Group | GSK1437173A _LD Group | GSK1437173A _MD Group | GSK1437173A _HD Group | Placebo + GSK1437173A _HD Group | GSK1437173A_MODIFIED Group
Number analyzed (Participants) | 100 | 102 | 108 | 97 | 33
T-cells/million cells
  Day 0: number analyzed (Participants) | 97 | 98 | 108 | 94 | 26
  Day 0 | 74.94 (113.07) | 87.33 (117.28) | 111.54 (204.36) | 81.54 (119.17) | 122.68 (362.64)
  Month 2: number analyzed (Participants) | 92 | 102 | 104 | 91 | 27
  Month 2 | 71.42 (96.41) | 83.01 (124.50) | 75.88 (129.33) | 111.15 (217.08) | 115.82 (356.29)
  Month 3: number analyzed (Participants) | 100 | 101 | 98 | 97 | 33
  Month 3 | 86.81 (120.39) | 76.75 (137.37) | 99.07 (139.42) | 106.97 (167.59) | 136.22 (470.58)

13. Secondary Outcome: Frequency of gE-specific CD8 T-cells Expressing CD40L and at Least Another Activation Marker
Description: Among other activation markers expressed were interleukin-2 [IL-2] or interferon-gamma [IFN-γ] or tumour necrosis factor-alpha [TNF-α]. Analysis of cytokines expression was done by means of in vitro flow cytometry using intracellular cytokine staining (ICS).
Time Frame: At pre-vaccination (Day 0), one month after the first vaccination (Month 2) and second vaccination (Month 3)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-cells/million cells
Arm/Group | GSK1437173A _LD Group | GSK1437173A _MD Group | GSK1437173A _HD Group | Placebo + GSK1437173A _HD Group | GSK1437173A_MODIFIED Group
Number analyzed (Participants) | 78 | 70 | 77 | 76 | 25
T-cells/million cells
  Day 0: number analyzed (Participants) | 65 | 70 | 77 | 67 | 23
  Day 0 | 41.35 (54.48) | 61.30 (118.43) | 56.85 (78.31) | 35.96 (69.51) | 59.94 (75.13)
  Month 2: number analyzed (Participants) | 62 | 70 | 63 | 69 | 25
  Month 2 | 63.87 (82.02) | 66.76 (90.29) | 47.20 (64.54) | 71.20 (93.18) | 54.63 (69.92)
  Month 3: number analyzed (Participants) | 78 | 69 | 74 | 76 | 23
  Month 3 | 69.50 (105.36) | 65.34 (64.17) | 85.57 (105.34) | 76.19 (72.44) | 33.12 (47.32)

14. Secondary Outcome: Anti-gE Specific Antibody Concentrations
Description: Concentrations were presented as geometric mean concentrations (GMCs) and expressed in enzyme-linked immunosorbent assay (ELISA) units per milliliter (EL.U/mL).
Time Frame: At pre-vaccination (Day 0), one month after the first vaccination (Month 2) and second vaccination (Month 3)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | GSK1437173A _LD Group | GSK1437173A _MD Group | GSK1437173A _HD Group | Placebo + GSK1437173A _HD Group | GSK1437173A_MODIFIED Group
Number analyzed (Participants) | 157 | 156 | 151 | 153 | 50
EL.U/mL
  Anti-gE, Day 0 | 351.6 [306.2 to 403.8] | 312.8 [268.1 to 365.0] | 416.1 [355.0 to 487.7] | 337.2 [285.8 to 397.7] | 323.7 [245.2 to 427.3]
  Anti-gE, Month 2 | 3667.6 [3158.6 to 4258.7] | 4139.4 [3443.8 to 4975.4] | 5485.6 [4657.2 to 6461.3] | 361.5 [304.6 to 429.0] | 2148.9 [1461.8 to 3158.9]
  Anti-gE, Month 3: number analyzed (Participants) | 155 | 156 | 151 | 153 | 49
  Anti-gE, Month 3 | 9315.3 [8283.2 to 10476.1] | 12898.0 [11681.2 to 14241.6] | 15626.5 [14030.3 to 17404.3] | 6287.2 [5372.0 to 7358.3] | 4298.3 [3220.0 to 5737.7]

15. Secondary Outcome: Anti-varicella Zoster Virus (VZV) Specific Antibody Concentrations
Description: Concentrations were presented as geometric mean concentrations (GMCs) and expressed in milli-international units per milliliter (mIU/mL), as assessed by ELISA.
Time Frame: At pre-vaccination (Day 0), one month after the first vaccination (Month 2) and second vaccination (Month 3)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | GSK1437173A _LD Group | GSK1437173A _MD Group | GSK1437173A _HD Group | Placebo + GSK1437173A _HD Group | GSK1437173A_MODIFIED Group
Number analyzed (Participants) | 157 | 156 | 151 | 153 | 50
mIU/mL
  Anti-VZV, Day 0 | 1334.9 [1181.9 to 1507.7] | 1212.0 [1063.9 to 1380.7] | 1510.7 [1336.4 to 1707.7] | 1356.3 [1184.9 to 1552.6] | 1422.5 [1153.4 to 1754.5]
  Anti-VZV, Month 2 | 4408.1 [3847.7 to 5050.1] | 5131.9 [4469.8 to 5892.0] | 6511.7 [5723.1 to 7409.0] | 1341.6 [1177.7 to 1528.3] | 3481.2 [2756.0 to 4397.3]
  Anti-VZV, Month 3: number analyzed (Participants) | 155 | 156 | 151 | 153 | 49
  Anti-VZV, Month 3 | 8821.6 [7959.3 to 9777.4] | 11451.0 [10507.9 to 12478.7] | 14143.5 [12876.9 to 15534.7] | 6432.2 [5591.8 to 7398.9] | 5357.6 [4297.3 to 6679.4]

16. Secondary Outcome: Frequency of gE-specific CD4/CD8 T-cells Expressing at Least Two Different Activation Markers
Description: Among the activation markers expressed were interleukin-2 [IL-2] and/or interferon-gamma [IFN-γ] and/or tumour necrosis factor-alpha [TNF-α] and/or cluster of differentiation 40-ligand [CD40-L]. Analysis of cytokines expression was done by means of in vitro flow cytometry using intracellular cytokine staining (ICS). Month 12, 24 and 36 CMI analyses on CD8+ T cells were not performed as no detectable CD8 T+ cell response was measured to any of the vaccine formulations in the primary (108494) study.
Time Frame: At Months 12, 24 and 36
Population: The analysis was performed on the Total cohort for persistence at Months 12, 24 and 36, which included all vaccinated subjects in the vaccination phase (Zoster-003) who were contacted at Months 12, 24 and 36 respectively.
Measure: Mean (Standard Deviation); unit: T-cells/million cells
Arm/Group | GSK1437173A _LD Group | GSK1437173A _MD Group | GSK1437173A _HD Group | Placebo + GSK1437173A _HD Group | GSK1437173A_MODIFIED Group
Number analyzed (Participants) | 150 | 148 | 151 | 151 | 45
T-cells/million cells
  CD4-All Doubles, Month 12: number analyzed (Participants) | 150 | 148 | 151 | 146 | 45
  CD4-All Doubles, Month 12 | 1135.8 (936.0) | 1275.5 (1195.4) | 1274.0 (995.0) | 340.4 (296.8) | 274.5 (217.3)
  CD4-All Doubles, Month 24: number analyzed (Participants) | 143 | 147 | 145 | 151 | 45
  CD4-All Doubles, Month 24 | 1004.1 (838.8) | 1195.5 (1375.5) | 1079.9 (948.0) | 244.1 (233.2) | 285.2 (255.6)
  CD4-All Doubles, Month 36: number analyzed (Participants) | 137 | 138 | 142 | 146 | 44
  CD4-All Doubles, Month 36 | 827.3 (922.9) | 969.7 (1034.9) | 896.3 (770.4) | 239.7 (181.7) | 229.7 (217.1)

17. Secondary Outcome: Frequency of gE-specific CD4/CD8 T-cells Expressing IFN-γ and at Least Another Activation Marker
Description: Among other activation markers expressed were interleukin-2 [IL-2] or tumour necrosis factor-alpha [TNF-α] or cluster of differentiation 40-ligand [CD40-L]. Analysis of cytokines expression was done by means of in vitro flow cytometry using intracellular cytokine staining (ICS). Month 12, 24 and 36 CMI analyses on CD8+ T cells were not performed as no detectable CD8 T+ cell response was measured to any of the vaccine formulations in the primary (108494) study.
Time Frame: At Months 12, 24 and 36
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: T-cells/million cells
Arm/Group | GSK1437173A _LD Group | GSK1437173A _MD Group | GSK1437173A _HD Group | Placebo + GSK1437173A _HD Group | GSK1437173A_MODIFIED Group
Number analyzed (Participants) | 150 | 148 | 151 | 151 | 45
T-cells/million cells
  Month 12: number analyzed (Participants) | 150 | 148 | 151 | 146 | 45
  Month 12 | 659.9 (594.3) | 767.8 (895.1) | 718.9 (634.2) | 235.5 (244.7) | 176.8 (152.7)
  Month 24: number analyzed (Participants) | 143 | 147 | 145 | 151 | 45
  Month 24 | 541.9 (503.1) | 668.9 (1140.6) | 543.6 (554.7) | 157.0 (183.4) | 181.2 (158.4)
  Month 36: number analyzed (Participants) | 137 | 138 | 142 | 146 | 44
  Month 36 | 491.8 (604.1) | 583.3 (819.0) | 492.3 (437.0) | 172.2 (155.1) | 162.0 (151.4)

18. Secondary Outcome: Frequency of gE-specific CD4/CD8 T-cells Expressing IL-2 and at Least Another Activation Marker
Description: Among other activation markers expressed were interferon-gamma [IFN-γ] or tumour necrosis factor-alpha [TNF-α] or cluster of differentiation 40-ligand [CD40-L]. Analysis of cytokines expression was done by means of in vitro flow cytometry using intracellular cytokine staining (ICS). Month 12, 24 and 36 CMI analyses on CD8+ T cells were not performed as no detectable CD8 T+ cell response was measured to any of the vaccine formulations in the primary (108494) study.
Time Frame: At Months 12, 24 and 36
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: T-cells/million cells
Arm/Group | GSK1437173A _LD Group | GSK1437173A _MD Group | GSK1437173A _HD Group | Placebo + GSK1437173A _HD Group | GSK1437173A_MODIFIED Group
Number analyzed (Participants) | 150 | 148 | 151 | 151 | 45
T-cells/million cells
  Month 12: number analyzed (Participants) | 150 | 148 | 151 | 146 | 45
  Month 12 | 1056.2 (901.0) | 1164.7 (1029.1) | 1168.3 (935.4) | 291.7 (266.6) | 243.9 (204.8)
  Month 24: number analyzed (Participants) | 143 | 147 | 145 | 151 | 45
  Month 24 | 943.0 (809.5) | 1100.2 (1158.9) | 1007.8 (909.5) | 213.0 (207.4) | 233.0 (244.5)
  Month 36: number analyzed (Participants) | 137 | 138 | 142 | 146 | 44
  Month 36 | 768.9 (871.5) | 890.2 (883.3) | 834.7 (743.9) | 205.8 (154.5) | 213.9 (202.2)

19. Secondary Outcome: Frequency of gE-specific CD4/CD8 T-cells Expressing TNFα and at Least Another Activation Marker
Description: Among other activation markers expressed were interleukin-2 [IL-2] or interferon-gamma [IFN-γ] or cluster of differentiation 40-ligand [CD40-L]. Analysis of cytokines expression was done by means of in vitro flow cytometry using intracellular cytokine staining (ICS). Month 12, 24 and 36 CMI analyses on CD8+ T cells were not performed as no detectable CD8 T+ cell response was measured to any of the vaccine formulations in the primary (108494) study.
Time Frame: At Month 12, 24 and 36
Population: as for outcome 16
Measure: Geometric Mean (Standard Deviation); unit: T-cells/million cells
Arm/Group | GSK1437173A _LD Group | GSK1437173A _MD Group | GSK1437173A _HD Group | Placebo + GSK1437173A _HD Group | GSK1437173A_MODIFIED Group
Number analyzed (Participants) | 150 | 148 | 151 | 151 | 45
T-cells/million cells
  Month 12: number analyzed (Participants) | 150 | 148 | 151 | 146 | 45
  Month 12 | 673.7 (616.0) | 736.2 (878.5) | 736.7 (660.7) | 193.2 (239.4) | 136.0 (132.8)
  Month 24: number analyzed (Participants) | 143 | 147 | 145 | 151 | 45
  Month 24 | 567.9 (527.7) | 663.1 (1097.0) | 591.5 (586.6) | 144.1 (196.1) | 133.0 (158.1)
  Month 36: number analyzed (Participants) | 137 | 138 | 142 | 146 | 44
  Month 36 | 497.4 (652.5) | 567.9 (808.4) | 510.7 (522.1) | 117.9 (151.7) | 98.1 (116.0)

20. Secondary Outcome: Frequency of gE-specific CD4/CD8 T-cells Expressing CD40L and at Least Another Activation Marker
Description: Among other activation markers expressed were interleukin-2 [IL-2] or interferon-gamma [IFN-γ] or tumour necrosis factor-alpha [TNF-α] . Analysis of cytokines expression was done by means of in vitro flow cytometry using intracellular cytokine staining (ICS). Month 12, 24 and 36 CMI analyses on CD8+ T cells were not performed as no detectable CD8 T+ cell response was measured to any of the vaccine formulations in the primary (108494) study.
Time Frame: At Month 12, 24 and 36
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: T-cells/million cells
Arm/Group | GSK1437173A _LD Group | GSK1437173A _MD Group | GSK1437173A _HD Group | Placebo + GSK1437173A _HD Group | GSK1437173A_MODIFIED Group
Number analyzed (Participants) | 150 | 148 | 151 | 151 | 45
T-cells/million cells
  Month 12: number analyzed (Participants) | 150 | 148 | 151 | 146 | 45
  Month 12 | 969.0 (811.8) | 1057.2 (943.4) | 1062.8 (850.3) | 267.5 (246.0) | 221.0 (180.9)
  Month 24: number analyzed (Participants) | 143 | 147 | 145 | 151 | 45
  Month 24 | 935.2 (801.5) | 1079.9 (1040.1) | 981.6 (890.9) | 210.8 (187.2) | 270.3 (248.6)
  Month 36: number analyzed (Participants) | 137 | 138 | 142 | 146 | 44
  Month 36 | 753.0 (852.9) | 912.9 (1009.2) | 823.0 (727.9) | 202.5 (166.3) | 202.8 (187.1)

21. Secondary Outcome: Anti-gE Specific Antibody Concentrations
Description: as for outcome 14
Time Frame: At Months 12, 24 and 36
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | GSK1437173A _LD Group | GSK1437173A _MD Group | GSK1437173A _HD Group | Placebo + GSK1437173A _HD Group | GSK1437173A_MODIFIED Group
Number analyzed (Participants) | 156 | 159 | 159 | 160 | 50
EL.U/mL
  Anti-gE, Month 12 | 3384.8 [2987.2 to 3835.4] | 4280.3 [3818.4 to 4798.0] | 5258.2 [4725.2 to 5851.3] | 1664.5 [1443.7 to 1919.1] | 1888.2 [1452.7 to 2454.1]
  Anti-gE, Month 24: number analyzed (Participants) | 149 | 155 | 154 | 157 | 48
  Anti-gE, Month 24 | 2363.8 [2081.0 to 2685.0] | 2784.6 [2494.0 to 3109.1] | 3390.0 [3013.6 to 3813.5] | 1126.3 [982.2 to 1291.6] | 1339.1 [1038.3 to 1727.0]
  Anti-gE, Month 36: number analyzed (Participants) | 146 | 146 | 150 | 152 | 47
  Anti-gE, Month 36 | 2064.1 [1834.6 to 2322.3] | 2444.3 [2175.2 to 2746.8] | 2956.4 [2653.6 to 3293.7] | 959.5 [831.0 to 1107.9] | 973.9 [755.4 to 1255.6]

22. Secondary Outcome: Anti-varicella Zoster Virus (VZV) Specific Antibody Concentrations
Description: Concentrations were presented as geometric mean concentrations (GMCs) and expressed in milli-international units per milliliter (mIU/mL).
Time Frame: At Months 12, 24 and 36
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | GSK1437173A _LD Group | GSK1437173A _MD Group | GSK1437173A _HD Group | Placebo + GSK1437173A _HD Group | GSK1437173A_MODIFIED Group
Number analyzed (Participants) | 149 | 155 | 154 | 157 | 48
mIU/mL
  Anti-VZV, Month 12: number analyzed (Participants) | 146 | 147 | 150 | 155 | 47
  Anti-VZV, Month 12 | 4190.1 [3845.4 to 4565.8] | 4761.3 [4367.0 to 5191.3] | 5559.1 [5141.5 to 6010.7] | 2704.1 [2424.5 to 3016.0] | 2733.8 [2208.8 to 3383.7]
  Anti-VZV, Month 24 | 2557.4 [2397.5 to 2727.8] | 2673.6 [2523.8 to 2832.3] | 2976.0 [2819.5 to 3141.3] | 1849.3 [1701.8 to 2009.5] | 1922.6 [1643.1 to 2249.6]
  Anti-VZV, Month 36: number analyzed (Participants) | 146 | 146 | 150 | 155 | 47
  Anti-VZV, Month 36 | 2426.6 [2257.2 to 2608.8] | 2555.0 [2385.8 to 2736.3] | 2826.7 [2648.4 to 3017.0] | 1729.9 [1582.5 to 1891.1] | 1739.9 [1481.0 to 2044.0]

23. Secondary Outcome: Frequency of VZV-specific Memory B-cells in a Subset of Subjects
Description: Memory B cells specific to the gE antigen, as assessed by the enzyme-linked immunosorbent spot (ELISPOT) method, were expressed as a frequency of the specific memory B-cells per million memory B-cells. Results were tabulated for subjects aged 70 years and older.
Time Frame: At pre-vaccination (Day 0) and at Month 3
Population: The analysis was performed on the Total cohort for persistence at Month 12, which included all vaccinated subjects in the vaccination phase (Zoster-003) who were contacted at Month 12.
Measure: Mean (Standard Deviation); unit: B-cells/million cells
Arm/Group | GSK1437173A _LD Group | GSK1437173A _MD Group | GSK1437173A _HD Group | Placebo + GSK1437173A _HD Group | GSK1437173A_MODIFIED Group
Number analyzed (Participants) | 19 | 23 | 23 | 21 | 8
B-cells/million cells
  Memory B-cells, Day 0: number analyzed (Participants) | 18 | 23 | 19 | 18 | 8
  Memory B-cells, Day 0 | 336.5 (359.5) | 490.4 (704.7) | 356.6 (348.0) | 332.3 (404.9) | 380.6 (299.7)
  Memory B-cells, Month 3: number analyzed (Participants) | 19 | 21 | 23 | 21 | 6
  Memory B-cells, Month 3 | 5699.3 (8166.2) | 5997.1 (5034.6) | 9707.5 (8787.1) | 1583.7 (2266.0) | 1042.2 (1139.9)

24. Secondary Outcome: Number of Subjects With Different Biochemical and Haematological Levels
Description: Among biochemical and haematological parameters assessed were albumin [ALB], alanine aminotransferase [ALT], aspartate aminotransferase [AST], basophils [BAS], calcium [CAL], eosinophils [EOS], fibrinogen [FIB], haematocrit [HEM], hemoglobin [Hgb], leucocytes [LEU], lymphocytes [LYM], lactate dehydrogenate [LDH], monocytes [MON], neutrophils [NEU], partial thromboplastin time [PTPT], platelets [PLA], pro thrombin time [PTT], red blood cells [RBC], serum creatinine [SCREA], total protein [TP]. Levels of haematological/biochemical parameters assessed in terms of normal laboratory values were - unknown, below, within and above.
Time Frame: At Day 0, Month 2 and Month 3
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with a least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A _LD Group | GSK1437173A _MD Group | GSK1437173A _HD Group | Placebo + GSK1437173A _HD Group | GSK1437173A_MODIFIED Group
Number analyzed (Participants) | 164 | 166 | 164 | 165 | 54
Participants
  ALB, Day 0: number analyzed (Participants) | 74 | 77 | 75 | 75 | 24
  ALB, Day 0: Unknown | 0 | 0 | 0 | 0 | 0
  ALB, Day 0: Below | 13 | 12 | 14 | 12 | 4
  ALB, Day 0: Within | 57 | 64 | 59 | 61 | 19
  ALB, Day 0: Above | 4 | 1 | 2 | 2 | 1
  ALB, Month 2: number analyzed (Participants) | 72 | 77 | 74 | 75 | 22
  ALB, Month 2: Unknown | 0 | 0 | 0 | 0 | 0
  ALB, Month 2: Below | 13 | 14 | 11 | 17 | 6
  ALB, Month 2: Within | 57 | 61 | 62 | 55 | 16
  ALB, Month 2: Above | 2 | 2 | 1 | 3 | 0
  ALB, Month 3: number analyzed (Participants) | 70 | 77 | 73 | 75 | 21
  ALB, Month 3: Unknown | 0 | 0 | 1 | 0 | 0
  ALB, Month 3: Below | 8 | 12 | 9 | 17 | 4
  ALB, Month 3: Within | 61 | 62 | 61 | 55 | 17
  ALB, Month 3: Above | 1 | 3 | 2 | 3 | 0
  ALT, Day 0: Unknown | 0 | 0 | 0 | 0 | 1
  ALT, Day 0: Below | 1 | 2 | 0 | 1 | 0
  ALT, Day 0: Within | 150 | 151 | 152 | 154 | 50
  ALT, Day 0: Above | 13 | 13 | 12 | 10 | 3
  ALT, Month 2: number analyzed (Participants) | 162 | 164 | 162 | 164 | 51
  ALT, Month 2: Unknown | 0 | 0 | 0 | 0 | 0
  ALT, Month 2: Below | 1 | 1 | 0 | 1 | 0
  ALT, Month 2: Within | 152 | 149 | 155 | 150 | 48
  ALT, Month 2: Above | 9 | 14 | 7 | 13 | 3
  ALT, Month 3: number analyzed (Participants) | 160 | 164 | 161 | 164 | 51
  ALT, Month 3: Unknown | 0 | 0 | 1 | 0 | 0
  ALT, Month 3: Below | 1 | 2 | 0 | 1 | 0
  ALT, Month 3: Within | 152 | 150 | 154 | 150 | 46
  ALT, Month 3: Above | 7 | 12 | 6 | 13 | 5
  AST, Day 0: Unknown | 0 | 0 | 0 | 0 | 0
  AST, Day 0: Below | 0 | 1 | 1 | 3 | 0
  AST, Day 0: Within | 156 | 154 | 156 | 148 | 51
  AST, Day 0: Above | 8 | 11 | 7 | 14 | 3
  AST, Month 2: number analyzed (Participants) | 162 | 164 | 162 | 164 | 51
  AST, Month 2: Unknown | 0 | 0 | 0 | 0 | 0
  AST, Month 2: Below | 0 | 1 | 0 | 0 | 0
  AST, Month 2: Within | 150 | 151 | 151 | 151 | 51
  AST, Month 2: Above | 12 | 12 | 11 | 13 | 0
  AST, Month 3: number analyzed (Participants) | 160 | 164 | 161 | 164 | 51
  AST, Month 3: Unknown | 0 | 0 | 2 | 0 | 0
  AST, Month 3: Below | 0 | 3 | 0 | 0 | 0
  AST, Month 3: Within | 151 | 146 | 153 | 153 | 48
  AST, Month 3: Above | 9 | 15 | 6 | 11 | 3
  BAS, Day 0: Unknown | 7 | 11 | 5 | 6 | 1
  BAS, Day 0: Below | 0 | 1 | 0 | 0 | 1
  BAS, Day 0: Within | 148 | 147 | 153 | 153 | 50
  BAS, Day 0: Above | 9 | 7 | 6 | 6 | 2
  BAS, Month 2: number analyzed (Participants) | 162 | 164 | 162 | 164 | 51
  BAS, Month 2: Unknown | 0 | 0 | 1 | 0 | 0
  BAS, Month 2: Below | 0 | 1 | 1 | 1 | 1
  BAS, Month 2: Within | 153 | 155 | 152 | 154 | 47
  BAS, Month 2: Above | 9 | 8 | 8 | 9 | 3
  BAS, Month 3: number analyzed (Participants) | 160 | 164 | 161 | 164 | 51
  BAS, Month 3: Unknown | 0 | 0 | 0 | 0 | 0
  BAS, Month 3: Below | 0 | 0 | 2 | 0 | 1
  BAS, Month 3: Within | 150 | 151 | 147 | 155 | 48
  BAS, Month 3: Above | 10 | 13 | 12 | 9 | 2
  CAL, Day 0: number analyzed (Participants) | 74 | 77 | 75 | 75 | 24
  CAL, Day 0: Unknown | 0 | 0 | 0 | 0 | 0
  CAL, Day 0: Below | 3 | 1 | 2 | 3 | 0
  CAL, Day 0: Within | 70 | 76 | 72 | 71 | 23
  CAL, Day 0: Above | 1 | 0 | 1 | 1 | 1
  CAL, Month 2: number analyzed (Participants) | 72 | 77 | 74 | 75 | 22
  CAL, Month 2: Unknown | 0 | 0 | 0 | 0 | 0
  CAL, Month 2: Below | 4 | 1 | 5 | 3 | 0
  CAL, Month 2: Within | 68 | 75 | 68 | 71 | 22
  CAL, Month 2: Above | 0 | 1 | 1 | 1 | 0
  CAL, Month 3: number analyzed (Participants) | 70 | 77 | 73 | 75 | 21
  CAL, Month 3: Unknown | 0 | 0 | 1 | 0 | 0
  CAL, Month 3: Below | 5 | 1 | 2 | 5 | 0
  CAL, Month 3: Within | 64 | 76 | 70 | 69 | 21
  CAL, Month 3: Above | 1 | 0 | 0 | 1 | 0
  EOS, Day 0: Unknown | 8 | 11 | 5 | 6 | 1
  EOS, Day 0: Below | 13 | 11 | 12 | 10 | 2
  EOS, Day 0: Within | 130 | 127 | 135 | 137 | 47
  EOS, Day 0: Above | 13 | 17 | 12 | 12 | 4
  EOS, Month 2: number analyzed (Participants) | 162 | 164 | 162 | 164 | 51
  EOS, Month 2: Unknown | 0 | 0 | 1 | 0 | 0
  EOS, Month 2: Below | 11 | 8 | 15 | 10 | 3
  EOS, Month 2: Within | 140 | 138 | 128 | 142 | 43
  EOS, Month 2: Above | 11 | 18 | 18 | 12 | 5
  EOS, Month 3: number analyzed (Participants) | 160 | 164 | 161 | 164 | 51
  EOS, Month 3: Unknown | 1 | 0 | 0 | 0 | 0
  EOS, Month 3: Below | 10 | 9 | 12 | 8 | 2
  EOS, Month 3: Within | 127 | 144 | 126 | 134 | 45
  EOS, Month 3: Above | 22 | 11 | 23 | 22 | 4
  FIB, Day 0: number analyzed (Participants) | 74 | 77 | 75 | 75 | 24
  FIB, Day 0: Unknown | 1 | 4 | 4 | 1 | 0
  FIB, Day 0: Below | 0 | 0 | 0 | 0 | 0
  FIB, Day 0: Within | 36 | 34 | 36 | 39 | 10
  FIB, Day 0: Above | 37 | 39 | 35 | 35 | 14
  FIB, Month 2: number analyzed (Participants) | 72 | 77 | 74 | 75 | 22
  FIB, Month 2: Unknown | 0 | 1 | 2 | 1 | 0
  FIB, Month 2: Below | 0 | 0 | 0 | 1 | 0
  FIB, Month 2: Within | 40 | 35 | 37 | 35 | 12
  FIB, Month 2: Above | 32 | 41 | 35 | 38 | 10
  FIB, Month 3: number analyzed (Participants) | 70 | 77 | 73 | 75 | 21
  FIB, Month 3: Unknown | 0 | 1 | 1 | 0 | 0
  FIB, Month 3: Below | 0 | 0 | 0 | 1 | 0
  FIB, Month 3: Within | 40 | 36 | 40 | 39 | 9
  FIB, Month 3: Above | 30 | 40 | 32 | 35 | 12
  HEM, Day 0: Unknown | 1 | 4 | 0 | 0 | 0
  HEM, Day 0: Below | 21 | 16 | 27 | 20 | 4
  HEM, Day 0: Within | 141 | 143 | 129 | 137 | 50
  HEM, Day 0: Above | 1 | 3 | 8 | 8 | 0
  HEM, Month 2: number analyzed (Participants) | 162 | 164 | 162 | 164 | 51
  HEM, Month 2: Unknown | 0 | 0 | 1 | 0 | 0
  HEM, Month 2: Below | 27 | 19 | 25 | 28 | 4
  HEM, Month 2: Within | 133 | 144 | 131 | 132 | 46
  HEM, Month 2: Above | 2 | 1 | 5 | 4 | 1
  HEM, Month 3: number analyzed (Participants) | 160 | 164 | 161 | 164 | 51
  HEM, Month 3: Unknown | 0 | 0 | 0 | 1 | 0
  HEM, Month 3: Below | 30 | 23 | 25 | 25 | 6
  HEM, Month 3: Within | 128 | 137 | 134 | 132 | 45
  HEM, Month 3: Above | 2 | 4 | 2 | 6 | 0
  HgB, Day 0: Unknown | 1 | 4 | 0 | 0 | 0
  HgB, Day 0: Below | 23 | 14 | 19 | 22 | 8
  HgB, Day 0: Within | 138 | 142 | 142 | 137 | 46
  HgB, Day 0: Above | 2 | 6 | 3 | 6 | 0
  HgB, Month 2: number analyzed (Participants) | 162 | 164 | 162 | 164 | 51
  HgB, Month 2: Unknown | 0 | 0 | 1 | 0 | 0
  HgB, Month 2: Below | 26 | 22 | 26 | 26 | 6
  HgB, Month 2: Within | 134 | 140 | 134 | 134 | 45
  HgB, Month 2: Above | 2 | 2 | 1 | 4 | 0
  HgB, Month 3: number analyzed (Participants) | 160 | 164 | 161 | 164 | 51
  HgB, Month 3: Unknown | 0 | 0 | 0 | 1 | 0
  HgB, Month 3: Below | 27 | 21 | 26 | 24 | 7
  HgB, Month 3: Within | 131 | 141 | 133 | 136 | 44
  HgB, Month 3: Above | 2 | 2 | 2 | 3 | 0
  LEU, Day 0: Unknown | 1 | 4 | 0 | 0 | 0
  LEU, Day 0: Below | 3 | 5 | 2 | 6 | 1
  LEU, Day 0: Within | 153 | 147 | 153 | 153 | 52
  LEU, Day 0: Above | 7 | 10 | 9 | 6 | 1
  LEU, Month 2: number analyzed (Participants) | 162 | 164 | 162 | 164 | 51
  LEU, Month 2: Unknown | 0 | 0 | 1 | 0 | 0
  LEU, Month 2: Below | 3 | 7 | 3 | 6 | 0
  LEU, Month 2: Within | 152 | 148 | 153 | 147 | 46
  LEU, Month 2: Above | 7 | 9 | 5 | 11 | 5
  LEU, Month 3: number analyzed (Participants) | 160 | 164 | 161 | 164 | 51
  LEU, Month 3: Unknown | 0 | 0 | 0 | 0 | 0
  LEU, Month 3: Below | 2 | 8 | 5 | 6 | 0
  LEU, Month 3: Within | 150 | 150 | 149 | 150 | 50
  LEU, Month 3: Above | 8 | 6 | 7 | 8 | 1
  LYM, Day 0: Unknown | 7 | 11 | 5 | 6 | 1
  LYM, Day 0: Below | 18 | 13 | 24 | 17 | 5
  LYM, Day 0: Within | 137 | 140 | 130 | 137 | 44
  LYM, Day 0: Above | 2 | 2 | 5 | 5 | 4
  LYM, Month 2: number analyzed (Participants) | 162 | 164 | 162 | 164 | 51
  LYM, Month 2: Unknown | 0 | 0 | 1 | 0 | 0
  LYM, Month 2: Below | 15 | 18 | 23 | 15 | 7
  LYM, Month 2: Within | 144 | 144 | 131 | 147 | 42
  LYM, Month 2: Above | 3 | 2 | 7 | 2 | 2
  LYM, Month 3: number analyzed (Participants) | 160 | 164 | 161 | 164 | 51
  LYM, Month 3: Unknown | 0 | 0 | 0 | 0 | 0
  LYM, Month 3: Below | 12 | 8 | 19 | 20 | 7
  LYM, Month 3: Within | 144 | 154 | 138 | 142 | 42
  LYM, Month 3: Above | 4 | 2 | 4 | 2 | 2
  LDH, Day 0: number analyzed (Participants) | 74 | 77 | 75 | 75 | 24
  LDH, Day 0: Unknown | 1 | 1 | 0 | 0 | 0
  LDH, Day 0: Below | 0 | 0 | 0 | 0 | 0
  LDH, Day 0: Within | 68 | 68 | 66 | 70 | 24
  LDH, Day 0: Above | 5 | 8 | 9 | 5 | 0
  LDH, Month 2: number analyzed (Participants) | 72 | 77 | 74 | 75 | 22
  LDH, Month 2: Unknown | 0 | 0 | 0 | 0 | 0
  LDH, Month 2: Below | 0 | 0 | 0 | 0 | 0
  LDH, Month 2: Within | 64 | 65 | 64 | 70 | 21
  LDH, Month 2: Above | 8 | 12 | 10 | 5 | 1
  LDH, Month 3: number analyzed (Participants) | 70 | 77 | 73 | 75 | 21
  LDH, Month 3: Unknown | 0 | 0 | 1 | 0 | 0
  LDH, Month 3: Below | 0 | 0 | 0 | 0 | 0
  LDH, Month 3: Within | 63 | 63 | 66 | 68 | 20
  LDH, Month 3: Above | 7 | 14 | 6 | 7 | 1
  MON, Day 0: Unknown | 7 | 11 | 5 | 6 | 1
  MON, Day 0: Below | 1 | 4 | 1 | 0 | 1
  MON, Day 0: Within | 148 | 142 | 147 | 148 | 49
  MON, Day 0: Above | 8 | 9 | 11 | 11 | 3
  MON, Month 2: number analyzed (Participants) | 162 | 164 | 162 | 164 | 51
  MON, Month 2: Unknown | 0 | 0 | 1 | 0 | 0
  MON, Month 2: Below | 0 | 0 | 2 | 0 | 0
  MON, Month 2: Within | 153 | 155 | 146 | 145 | 48
  MON, Month 2: Above | 9 | 9 | 13 | 19 | 3
  MON, Month 3: number analyzed (Participants) | 160 | 164 | 161 | 164 | 51
  MON, Month 3: Unknown | 0 | 0 | 0 | 0 | 0
  MON, Month 3: Below | 2 | 1 | 1 | 3 | 0
  MON, Month 3: Within | 145 | 151 | 145 | 148 | 49
  MON, Month 3: Above | 13 | 12 | 15 | 13 | 2
  NEU, Day 0: Unknown | 8 | 11 | 5 | 6 | 1
  NEU, Day 0: Below | 3 | 2 | 3 | 3 | 3
  NEU, Day 0: Within | 145 | 141 | 147 | 146 | 48
  NEU, Day 0: Above | 8 | 12 | 9 | 10 | 2
  NEU, Month 2: number analyzed (Participants) | 162 | 164 | 162 | 164 | 51
  NEU, Month 2: Unknown | 1 | 0 | 1 | 0 | 0
  NEU, Month 2: Below | 2 | 5 | 4 | 6 | 1
  NEU, Month 2: Within | 150 | 152 | 144 | 151 | 47
  NEU, Month 2: Above | 9 | 7 | 13 | 7 | 3
  NEU, Month 3: number analyzed (Participants) | 160 | 164 | 161 | 164 | 51
  NEU, Month 3: Unknown | 1 | 0 | 0 | 0 | 0
  NEU, Month 3: Below | 7 | 3 | 7 | 6 | 2
  NEU, Month 3: Within | 146 | 157 | 145 | 149 | 46
  NEU, Month 3: Above | 6 | 4 | 9 | 9 | 3
  PTPT, Day 0: number analyzed (Participants) | 53 | 55 | 53 | 51 | 16
  PTPT, Day 0: Unknown | 3 | 4 | 3 | 0 | 0
  PTPT, Day 0: Below | 5 | 2 | 2 | 3 | 0
  PTPT, Day 0: Within | 42 | 42 | 42 | 43 | 11
  PTPT, Day 0: Above | 3 | 7 | 6 | 5 | 5
  PTPT, Month 2: number analyzed (Participants) | 72 | 74 | 72 | 74 | 22
  PTPT, Month 2: Unknown | 0 | 1 | 3 | 1 | 0
  PTPT, Month 2: Below | 7 | 4 | 6 | 3 | 0
  PTPT, Month 2: Within | 59 | 58 | 57 | 64 | 20
  PTPT, Month 2: Above | 6 | 11 | 6 | 6 | 2
  PTPT, Month 3: number analyzed (Participants) | 70 | 77 | 73 | 75 | 21
  PTPT, Month 3: Unknown | 0 | 0 | 1 | 0 | 0
  PTPT, Month 3: Below | 4 | 4 | 6 | 5 | 1
  PTPT, Month 3: Within | 62 | 61 | 59 | 62 | 18
  PTPT, Month 3: Above | 4 | 12 | 7 | 8 | 2
  PLA, Day 0: Unknown | 1 | 4 | 0 | 0 | 0
  PLA, Day 0: Below | 6 | 4 | 9 | 10 | 2
  PLA, Day 0: Within | 147 | 150 | 149 | 148 | 49
  PLA, Day 0: Above | 10 | 8 | 6 | 7 | 3
  PLA, Month 2: number analyzed (Participants) | 162 | 164 | 162 | 164 | 51
  PLA, Month 2: Unknown | 0 | 0 | 1 | 0 | 0
  PLA, Month 2: Below | 6 | 7 | 11 | 12 | 1
  PLA, Month 2: Within | 150 | 152 | 145 | 145 | 49
  PLA, Month 2: Above | 6 | 5 | 5 | 7 | 1
  PLA, Month 3: number analyzed (Participants) | 160 | 164 | 161 | 164 | 51
  PLA, Month 3: Unknown | 0 | 0 | 0 | 1 | 0
  PLA, Month 3: Below | 6 | 6 | 9 | 12 | 3
  PLA, Month 3: Within | 149 | 153 | 147 | 148 | 46
  PLA, Month 3: Above | 5 | 5 | 5 | 3 | 2
  PTT, Day 0: number analyzed (Participants) | 53 | 55 | 53 | 51 | 16
  PTT, Day 0: Unknown | 3 | 3 | 3 | 0 | 0
  PTT, Day 0: Below | 4 | 9 | 5 | 5 | 5
  PTT, Day 0: Within | 44 | 38 | 42 | 44 | 11
  PTT, Day 0: Above | 2 | 5 | 3 | 2 | 0
  PTT, Month 2: number analyzed (Participants) | 72 | 74 | 72 | 74 | 22
  PTT, Month 2: Unknown | 0 | 1 | 3 | 1 | 0
  PTT, Month 2: Below | 5 | 10 | 6 | 7 | 3
  PTT, Month 2: Within | 65 | 62 | 61 | 65 | 19
  PTT, Month 2: Above | 2 | 1 | 2 | 1 | 0
  PTT, Month 3: number analyzed (Participants) | 70 | 77 | 73 | 75 | 21
  PTT, Month 3: Unknown | 0 | 0 | 1 | 0 | 0
  PTT, Month 3: Below | 5 | 10 | 6 | 8 | 2
  PTT, Month 3: Within | 62 | 64 | 63 | 64 | 19
  PTT, Month 3: Above | 3 | 3 | 3 | 3 | 0
  RBC, Day 0: Unknown | 1 | 5 | 2 | 1 | 0
  RBC, Day 0: Below | 23 | 21 | 25 | 23 | 9
  RBC, Day 0: Within | 137 | 135 | 128 | 136 | 42
  RBC, Day 0: Above | 3 | 5 | 9 | 5 | 3
  RBC, Month 2: number analyzed (Participants) | 162 | 164 | 162 | 164 | 51
  RBC, Month 2: Unknown | 0 | 1 | 1 | 0 | 0
  RBC, Month 2: Below | 25 | 23 | 27 | 24 | 8
  RBC, Month 2: Within | 136 | 138 | 128 | 135 | 42
  RBC, Month 2: Above | 1 | 2 | 6 | 5 | 1
  RBC, Month 3: number analyzed (Participants) | 160 | 164 | 161 | 164 | 51
  RBC, Month 3: Unknown | 1 | 0 | 0 | 1 | 0
  RBC, Month 3: Below | 27 | 23 | 26 | 23 | 5
  RBC, Month 3: Within | 129 | 138 | 131 | 136 | 46
  RBC, Month 3: Above | 3 | 3 | 4 | 4 | 0
  SCREA, Day 0: Unknown | 1 | 1 | 1 | 0 | 0
  SCREA, Day 0: Below | 4 | 2 | 3 | 3 | 0
  SCREA, Day 0: Within | 130 | 132 | 128 | 135 | 43
  SCREA, Day 0: Above | 29 | 31 | 32 | 27 | 11
  SCREA, Month 2: number analyzed (Participants) | 162 | 164 | 162 | 164 | 51
  SCREA, Month 2: Unknown | 0 | 0 | 0 | 0 | 0
  SCREA, Month 2: Below | 3 | 2 | 1 | 3 | 2
  SCREA, Month 2: Within | 135 | 131 | 129 | 131 | 38
  SCREA, Month 2: Above | 24 | 31 | 32 | 30 | 11
  SCREA, Month 3: number analyzed (Participants) | 160 | 164 | 161 | 164 | 51
  SCREA, Month 3: Unknown | 0 | 0 | 1 | 0 | 0
  SCREA, Month 3: Below | 3 | 3 | 2 | 2 | 0
  SCREA, Month 3: Within | 132 | 127 | 130 | 134 | 42
  SCREA, Month 3: Above | 25 | 34 | 28 | 28 | 9
  TP, Day 0: number analyzed (Participants) | 74 | 77 | 75 | 75 | 24
  TP, Day 0: Unknown | 0 | 0 | 0 | 0 | 0
  TP, Day 0: Below | 6 | 2 | 9 | 3 | 1
  TP, Day 0: Within | 68 | 75 | 66 | 72 | 23
  TP, Day 0: Above | 0 | 0 | 0 | 0 | 0
  TP, Month 2: number analyzed (Participants) | 72 | 77 | 74 | 75 | 22
  TP, Month 2: Unknown | 0 | 0 | 0 | 0 | 0
  TP, Month 2: Below | 6 | 2 | 9 | 4 | 2
  TP, Month 2: Within | 66 | 75 | 65 | 71 | 20
  TP, Month 2: Above | 0 | 0 | 0 | 0 | 0
  TP, Month 3: number analyzed (Participants) | 70 | 77 | 73 | 75 | 21
  TP, Month 3: Unknown | 0 | 0 | 1 | 0 | 0
  TP, Month 3: Below | 3 | 7 | 13 | 6 | 0
  TP, Month 3: Within | 67 | 70 | 58 | 69 | 21
  TP, Month 3: Above | 0 | 0 | 1 | 0 | 0

25. Secondary Outcome: Number of German Subjects With Different Biochemical and Haematological Levels
Description: Among biochemical and haematological parameters assessed were albumin [ALB], calcium [CAL], fibrinogen [FIB], lactate dehydrogenase [LDH], partial thrombo-plastin time [PTPT], pro thrombin time [PTT], total protein [TP]. Levels of haematological/biochemical parameters assessed in terms of normal laboratory values were - below, within, above and missing, as compared to the pre-vaccination status (below, within, above or missing). Values for electrophoresis (globulins and albumin/globulin ratio) were not displayed.
Time Frame: At one week post-vaccination 1 (Month 0)
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A _LD Group | GSK1437173A _MD Group | GSK1437173A _HD Group | Placebo + GSK1437173A _HD Group | GSK1437173A_MODIFIED Group
Number analyzed (Participants) | 22 | 24 | 24 | 24 | 8
Participants
  ALB - Below: number analyzed (Participants) | 8 | 7 | 10 | 7 | 2
  ALB - Below: Below | 8 | 7 | 10 | 7 | 2
  ALB - Below: Within | 0 | 0 | 0 | 0 | 0
  ALB - Below: Above | 0 | 0 | 0 | 0 | 0
  ALB - Below: Missing | 0 | 0 | 0 | 0 | 0
  ALB - Within: number analyzed (Participants) | 16 | 17 | 14 | 17 | 6
  ALB - Within: Below | 3 | 5 | 2 | 4 | 2
  ALB - Within: Within | 12 | 12 | 12 | 12 | 4
  ALB - Within: Above | 0 | 0 | 0 | 0 | 0
  ALB - Within: Missing | 1 | 0 | 0 | 1 | 0
  CAL - Below: number analyzed (Participants) | 2 | 1 | 0 | 0 | 0
  CAL - Below: Below | 1 | 1 |  |  |
  CAL - Below: Within | 1 | 0 |  |  |
  CAL - Below: Above | 0 | 0 |  |  |
  CAL - Below: Missing | 0 | 0 |  |  |
  CAL - Within: number analyzed (Participants) | 21 | 23 | 24 | 24 | 8
  CAL - Within: Below | 1 | 0 | 1 | 0 | 0
  CAL - Within: Within | 19 | 23 | 21 | 22 | 8
  CAL - Within: Above | 0 | 0 | 2 | 1 | 0
  CAL - Within: Missing | 1 | 0 | 0 | 1 | 0
  CAL - Above: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  CAL - Above: Below | 0 |  |  |  |
  CAL - Above: Within | 1 |  |  |  |
  CAL - Above: Above | 0 |  |  |  |
  CAL - Above: Missing | 0 |  |  |  |
  FIB - Within: number analyzed (Participants) | 15 | 13 | 12 | 16 | 5
  FIB - Within: Below | 0 | 0 | 0 | 0 | 0
  FIB - Within: Within | 9 | 5 | 8 | 13 | 4
  FIB - Within: Above | 6 | 8 | 4 | 3 | 1
  FIB - Within: Missing | 0 | 0 | 0 | 0 | 0
  FIB - Above: number analyzed (Participants) | 9 | 11 | 12 | 8 | 3
  FIB - Above: Below | 0 | 0 | 0 | 0 | 0
  FIB - Above: Within | 0 | 0 | 2 | 3 | 0
  FIB - Above: Above | 8 | 11 | 10 | 4 | 3
  FIB - Above: Missing | 1 | 0 | 0 | 1 | 0
  LDH- Within: number analyzed (Participants) | 21 | 19 | 20 | 23 | 8
  LDH- Within: Below | 0 | 0 | 0 | 0 | 0
  LDH- Within: Within | 18 | 19 | 19 | 22 | 8
  LDH- Within: Above | 2 | 0 | 1 | 0 | 0
  LDH- Within: Missing | 1 | 0 | 0 | 1 | 0
  LDH- Above: number analyzed (Participants) | 2 | 5 | 4 | 1 | 0
  LDH- Above: Below | 0 | 0 | 0 | 0 |
  LDH- Above: Within | 1 | 3 | 1 | 1 |
  LDH- Above: Above | 1 | 2 | 3 | 0 |
  LDH- Above: Missing | 0 | 0 | 0 | 0 |
  LDH- Missing: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  LDH- Missing: Below | 0 |  |  |  |
  LDH- Missing: Within | 0 |  |  |  |
  LDH- Missing: Above | 1 |  |  |  |
  LDH- Missing: Missing | 0 |  |  |  |
  PTPT - Missing: number analyzed (Participants) | 22 | 24 | 23 | 24 | 8
  PTPT - Missing: Below | 0 | 0 | 0 | 0 | 0
  PTPT - Missing: Within | 0 | 0 | 0 | 0 | 0
  PTPT - Missing: Above | 0 | 0 | 0 | 0 | 0
  PTPT - Missing: Missing | 22 | 24 | 23 | 24 | 8
  PTT - Missing: number analyzed (Participants) | 22 | 24 | 23 | 24 | 8
  PTT - Missing: Below | 0 | 0 | 0 | 0 | 0
  PTT - Missing: Within | 0 | 0 | 0 | 0 | 0
  PTT - Missing: Above | 0 | 0 | 1 | 0 | 0
  PTT - Missing: Missing | 22 | 24 | 22 | 24 | 8
  TP - Below: number analyzed (Participants) | 2 | 0 | 1 | 0 | 0
  TP - Below: Below | 0 |  | 0 |  |
  TP - Below: Within | 2 |  | 1 |  |
  TP - Below: Above | 0 |  | 0 |  |
  TP - Below: Missing | 0 |  | 0 |  |
  TP - Within: number analyzed (Participants) | 22 | 24 | 23 | 24 | 8
  TP - Within: Below | 0 | 0 | 2 | 1 | 0
  TP - Within: Within | 21 | 24 | 21 | 22 | 8
  TP - Within: Above | 0 | 0 | 0 | 0 | 0
  TP - Within: Missing | 1 | 0 | 0 | 1 | 0

26. Secondary Outcome: Number of German Subjects With Different Biochemical and Haematological Levels
Description: as for outcome 25
Time Frame: At one week post-vaccination 2 (Month 2)
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A _LD Group | GSK1437173A _MD Group | GSK1437173A _HD Group | Placebo + GSK1437173A _HD Group | GSK1437173A_MODIFIED Group
Number analyzed (Participants) | 22 | 24 | 24 | 24 | 8
Participants
  ALB - Below: number analyzed (Participants) | 8 | 7 | 10 | 7 | 2
  ALB - Below: Below | 4 | 6 | 8 | 6 | 2
  ALB - Below: Within | 1 | 1 | 1 | 0 | 0
  ALB - Below: Above | 0 | 0 | 0 | 0 | 0
  ALB - Below: Missing | 3 | 0 | 1 | 1 | 0
  ALB - Within: number analyzed (Participants) | 16 | 17 | 14 | 17 | 6
  ALB - Within: Below | 2 | 2 | 2 | 4 | 1
  ALB - Within: Within | 12 | 15 | 11 | 12 | 5
  ALB - Within: Above | 0 | 0 | 0 | 0 | 0
  ALB - Within: Missing | 2 | 0 | 1 | 1 | 0
  CAL - Below: number analyzed (Participants) | 2 | 1 | 0 | 0 | 0
  CAL - Below: Below | 1 | 0 |  |  |
  CAL - Below: Within | 0 | 1 |  |  |
  CAL - Below: Above | 0 | 0 |  |  |
  CAL - Below: Missing | 1 | 0 |  |  |
  CAL - Within: number analyzed (Participants) | 21 | 23 | 24 | 24 | 8
  CAL - Within: Below | 0 | 0 | 2 | 0 | 0
  CAL - Within: Within | 16 | 23 | 20 | 22 | 8
  CAL - Within: Above | 1 | 0 | 0 | 0 | 0
  CAL - Within: Missing | 4 | 0 | 2 | 2 | 0
  CAL - Above: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  CAL - Above: Below | 0 |  |  |  |
  CAL - Above: Within | 1 |  |  |  |
  CAL - Above: Above | 0 |  |  |  |
  CAL - Above: Missing | 0 |  |  |  |
  FIB - Within: number analyzed (Participants) | 15 | 13 | 12 | 16 | 5
  FIB - Within: Below | 0 | 0 | 0 | 0 | 0
  FIB - Within: Within | 8 | 8 | 6 | 11 | 4
  FIB - Within: Above | 5 | 5 | 5 | 3 | 1
  FIB - Within: Missing | 2 | 0 | 1 | 2 | 0
  FIB - Above: number analyzed (Participants) | 9 | 11 | 12 | 8 | 3
  FIB - Above: Below | 0 | 0 | 0 | 0 | 0
  FIB - Above: Within | 0 | 1 | 3 | 1 | 0
  FIB - Above: Above | 6 | 10 | 8 | 7 | 3
  FIB - Above: Missing | 3 | 0 | 1 | 0 | 0
  LDH - Within: number analyzed (Participants) | 21 | 19 | 20 | 23 | 8
  LDH - Within: Below | 0 | 0 | 0 | 0 | 0
  LDH - Within: Within | 14 | 16 | 15 | 20 | 8
  LDH - Within: Above | 2 | 3 | 3 | 1 | 0
  LDH - Within: Missing | 5 | 0 | 2 | 2 | 0
  LDH - Above: number analyzed (Participants) | 2 | 5 | 4 | 1 | 0
  LDH - Above: Below | 0 | 0 | 0 | 0 |
  LDH - Above: Within | 0 | 4 | 1 | 1 |
  LDH - Above: Above | 2 | 1 | 3 | 0 |
  LDH - Above: Missing | 0 | 0 | 0 | 0 |
  LDH - Missing: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  LDH - Missing: Below | 0 |  |  |  |
  LDH - Missing: Within | 1 |  |  |  |
  LDH - Missing: Above | 0 |  |  |  |
  LDH - Missing: Missing | 0 |  |  |  |
  PTPT - Missing: number analyzed (Participants) | 22 | 24 | 23 | 24 | 8
  PTPT - Missing: Below | 0 | 1 | 2 | 1 | 0
  PTPT - Missing: Within | 18 | 22 | 20 | 19 | 8
  PTPT - Missing: Above | 1 | 1 | 0 | 2 | 0
  PTPT - Missing: Missing | 3 | 0 | 1 | 2 | 0
  PTT - Missing: number analyzed (Participants) | 22 | 24 | 23 | 24 | 8
  PTT - Missing: Below | 1 | 1 | 0 | 2 | 0
  PTT - Missing: Within | 18 | 23 | 22 | 20 | 8
  PTT - Missing: Above | 0 | 0 | 0 | 0 | 0
  PTT - Missing: Missing | 3 | 0 | 1 | 2 | 0
  TP - Below: number analyzed (Participants) | 2 | 0 | 1 | 0 | 0
  TP - Below: Below | 0 |  | 0 |  |
  TP - Below: Within | 0 |  | 1 |  |
  TP - Below: Above | 0 |  | 0 |  |
  TP - Below: Missing | 2 |  | 0 |  |
  TP - Within: number analyzed (Participants) | 22 | 24 | 23 | 24 | 8
  TP - Within: Below | 0 | 0 | 2 | 2 | 0
  TP - Within: Within | 19 | 24 | 19 | 20 | 8
  TP - Within: Above | 0 | 0 | 0 | 0 | 0
  TP - Within: Missing | 3 | 0 | 2 | 2 | 0

27. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with a least one vaccine administration documented, who filled in their symptom sheets.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A _LD Group | GSK1437173A _MD Group | GSK1437173A _HD Group | Placebo + GSK1437173A _HD Group | GSK1437173A_MODIFIED Group
Number analyzed (Participants) | 164 | 166 | 165 | 165 | 54
Participants
  Any Pain, Dose 1 | 94 | 11 | 99 | 2 | 7
  Grade 3 Pain, Dose 1 | 0 | 0 | 3 | 0 | 0
  Any Redness, Dose 1 | 40 | 49 | 43 | 1 | 2
  Grade 3 Redness, Dose 1 | 2 | 2 | 3 | 0 | 0
  Any Swelling, Dose 1 | 26 | 21 | 24 | 3 | 1
  Grade 3 Swelling, Dose 1 | 1 | 2 | 2 | 0 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 159 | 164 | 161 | 163 | 51
  Any Pain, Dose 2 | 99 | 93 | 99 | 93 | 4
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 159 | 164 | 161 | 163 | 51
  Grade 3 Pain, Dose 2 | 4 | 3 | 3 | 3 | 0
  Any Redness, Dose 2: number analyzed (Participants) | 159 | 164 | 161 | 163 | 51
  Any Redness, Dose 2 | 51 | 54 | 52 | 48 | 2
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 159 | 164 | 161 | 163 | 51
  Grade 3 Redness, Dose 2 | 1 | 3 | 2 | 2 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 159 | 164 | 161 | 163 | 51
  Any Swelling, Dose 2 | 30 | 23 | 30 | 27 | 0
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 159 | 164 | 161 | 163 | 51
  Grade 3 Swelling, Dose 2 | 0 | 0 | 1 | 0 | 0
  Any Pain, Across doses | 115 | 12 | 122 | 93 | 9
  Grade 3 Pain, Across doses | 4 | 3 | 6 | 3 | 0
  Any Redness, Across doses | 68 | 66 | 68 | 49 | 2
  Grade 3 Redness, Across doses | 2 | 5 | 4 | 2 | 0
  Any Swelling, Across doses | 44 | 33 | 45 | 30 | 1
  Grade 3 Swelling, Across doses | 1 | 2 | 2 | 0 | 0

28. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were arthralgia, fatigue, fever [defined as oral temperature equal to or above (≥) 37.5 degrees Celsius (°C)], headache and myalgia. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A _LD Group | GSK1437173A _MD Group | GSK1437173A _HD Group | Placebo + GSK1437173A _HD Group | GSK1437173A_MODIFIED Group
Number analyzed (Participants) | 164 | 166 | 165 | 165 | 54
Participants
  Any Fatigue, Dose 1 | 36 | 48 | 46 | 20 | 8
  Grade 3 Fatigue, Dose 1 | 1 | 2 | 2 | 2 | 1
  Related Fatigue, Dose 1 | 30 | 34 | 34 | 12 | 6
  Any Fever, Dose 1 | 7 | 7 | 5 | 4 | 0
  Grade 3 Fever, Dose 1 | 0 | 0 | 0 | 0 | 0
  Related Fever, Dose 1 | 7 | 5 | 3 | 4 | 0
  Any Headache, Dose 1 | 23 | 25 | 24 | 13 | 7
  Grade 3 Headache, Dose 1 | 0 | 0 | 2 | 0 | 0
  Related Headache, Dose 1 | 19 | 17 | 13 | 6 | 6
  Any Myalgia, Dose 1 | 48 | 57 | 46 | 11 | 8
  Grade 3 Myalgia, Dose 1 | 1 | 2 | 2 | 1 | 0
  Related Myalgia, Dose 1 | 41 | 52 | 41 | 10 | 6
  Any Fatigue, Dose 2: number analyzed (Participants) | 159 | 164 | 161 | 163 | 51
  Any Fatigue, Dose 2 | 56 | 70 | 52 | 38 | 9
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 159 | 164 | 161 | 163 | 51
  Grade 3 Fatigue, Dose 2 | 2 | 6 | 4 | 1 | 0
  Related Fatigue, Dose 2: number analyzed (Participants) | 159 | 164 | 161 | 163 | 51
  Related Fatigue, Dose 2 | 47 | 48 | 43 | 27 | 7
  Any Fever, Dose 2: number analyzed (Participants) | 159 | 164 | 161 | 163 | 51
  Any Fever, Dose 2 | 13 | 13 | 18 | 5 | 0
  Grade 3 Fever, Dose 2: number analyzed (Participants) | 159 | 164 | 161 | 163 | 51
  Grade 3 Fever, Dose 2 | 0 | 1 | 0 | 0 | 0
  Related Fever, Dose 2: number analyzed (Participants) | 159 | 164 | 161 | 163 | 51
  Related Fever, Dose 2 | 12 | 12 | 18 | 5 | 0
  Any Headache, Dose 2: number analyzed (Participants) | 159 | 164 | 161 | 163 | 51
  Any Headache, Dose 2 | 39 | 47 | 39 | 27 | 7
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 159 | 164 | 161 | 163 | 51
  Grade 3 Headache, Dose 2 | 2 | 3 | 2 | 0 | 0
  Related Headache, Dose 2: number analyzed (Participants) | 159 | 164 | 161 | 163 | 51
  Related Headache, Dose 2 | 32 | 32 | 35 | 21 | 5
  Any Myalgia, Dose 2: number analyzed (Participants) | 159 | 164 | 161 | 163 | 51
  Any Myalgia, Dose 2 | 59 | 71 | 59 | 46 | 5
  Grade 3 Myalgia, Dose 2: number analyzed (Participants) | 159 | 164 | 161 | 163 | 51
  Grade 3 Myalgia, Dose 2 | 4 | 7 | 4 | 2 | 0
  Related Myalgia, Dose 2: number analyzed (Participants) | 159 | 164 | 161 | 163 | 51
  Related Myalgia, Dose 2 | 52 | 61 | 57 | 41 | 4
  Any Fatigue, Across doses | 69 | 85 | 73 | 47 | 1
  Grade 3 Fatigue, Across doses | 3 | 7 | 6 | 3 | 1
  Related Fatigue, Across doses | 57 | 60 | 59 | 33 | 9
  Any Fever, Across doses | 19 | 18 | 22 | 9 | 0
  Grade 3 Fever, Across doses | 0 | 1 | 0 | 0 | 0
  Related Fever, Across doses | 18 | 15 | 20 | 9 | 0
  Any Headache, Across doses | 47 | 59 | 51 | 36 | 9
  Grade 3 Headache, Across doses | 2 | 3 | 4 | 0 | 0
  Related Headache, Across doses | 39 | 41 | 42 | 25 | 7
  Any Myalgia, Across doses | 74 | 89 | 70 | 49 | 9
  Grade 3 Myalgia, Across doses | 5 | 8 | 6 | 3 | 0
  Related Myalgia, Across doses | 66 | 80 | 67 | 46 | 7

29. Secondary Outcome: Number of Subjects With Occurrence of Clinically Diagnosed Herpes Zoster (HZ) Episodes
Description: Clinically diagnosed episodes included rash that was assessed by hives, idiopathic thrombocytopenic purpura, petechiae.
Time Frame: From Month 0 to Month 3
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A _LD Group | GSK1437173A _MD Group | GSK1437173A _HD Group | Placebo + GSK1437173A _HD Group | GSK1437173A_MODIFIED Group
Number analyzed (Participants) | 164 | 166 | 165 | 165 | 54
Participants | 1 | 0 | 0 | 0 | 0

30. Secondary Outcome: Number of Subjects With Occurrence of Clinically Diagnosed HZ Episodes
Description: Clinically diagnosed episodes included rash that was assessed by hives, idiopathic thrombocytopenic purpura, petechiae.
Time Frame: From Month 3 up to Month 36
Population: The analysis was performed on the Total cohort for persistence at Months 12, 24 and 36, which included all vaccinated subjects in the vaccination phase (Zoster-003) who were contacted at Months 12, 24 and 36.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A _LD Group | GSK1437173A _MD Group | GSK1437173A _HD Group | Placebo + GSK1437173A _HD Group | GSK1437173A_MODIFIED Group
Number analyzed (Participants) | 156 | 159 | 159 | 161 | 50
Participants
  Month 3 - Month 12 | 0 | 0 | 0 | 1 | 0
  Month 12 - Month 24: number analyzed (Participants) | 150 | 155 | 154 | 157 | 49
  Month 12 - Month 24 | 1 | 0 | 0 | 0 | 0
  Month 24 - Month 36: number analyzed (Participants) | 147 | 147 | 150 | 155 | 47
  Month 24 - Month 36 | 0 | 0 | 0 | 0 | 1

31. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: During the 30-day (Days 0-29) post-vaccination period
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A _LD Group | GSK1437173A _MD Group | GSK1437173A _HD Group | Placebo + GSK1437173A _HD Group | GSK1437173A_MODIFIED Group
Number analyzed (Participants) | 164 | 166 | 165 | 165 | 54
Participants
  Any AE(s) | 55 | 52 | 54 | 41 | 16
  Grade 3 AE(s) | 7 | 10 | 10 | 5 | 4
  Related AE(s) | 20 | 22 | 24 | 13 | 2

32. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From Month 0 to Month 3
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A _LD Group | GSK1437173A _MD Group | GSK1437173A _HD Group | Placebo + GSK1437173A _HD Group | GSK1437173A_MODIFIED Group
Number analyzed (Participants) | 164 | 166 | 165 | 165 | 54
Participants | 2 | 4 | 3 | 6 | 3

33. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: as for outcome 32
Time Frame: From Month 3 to Month 12
Population: as for outcome 30
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A _LD Group | GSK1437173A _MD Group | GSK1437173A _HD Group | Placebo + GSK1437173A _HD Group | GSK1437173A_MODIFIED Group
Number analyzed (Participants) | 156 | 159 | 159 | 161 | 50
Participants
  Month 3 - Month 12 | 11 | 14 | 11 | 16 | 3
  Month 12 - Month 24: number analyzed (Participants) | 150 | 155 | 154 | 157 | 49
  Month 12 - Month 24 | 21 | 27 | 29 | 25 | 11
  Month 24 - Month 36: number analyzed (Participants) | 147 | 147 | 150 | 155 | 47
  Month 24 - Month 36 | 19 | 12 | 25 | 20 | 5

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 7-day (Days 0-6) post-vaccination period; Unsolicited AEs: during the 30-day (Days 0-29) post-vaccination period; SAEs: during the entire study period (from Day 0 to Month 36).
Groups:
- Placebo Group: Healthy male or female subjects aged 60 years or older, who received 2 doses of GSK1437173A modified formulation vaccine reconstituted with saline solution, according to a 0, 2-month schedule. The vaccine was administrated by (IM) in the upper deltoid site of the left arm.
Arm/Group | GSK1437173A _LD Group | GSK1437173A _MD Group | GSK1437173A _HD Group | Placebo + GSK1437173A _HD Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 2/164 | 3/166 | 3/165 | 5/165 | 1/54
Serious Adverse Events (participants affected / at risk) | 53/164 | 57/166 | 68/165 | 67/165 | 22/54
Other Adverse Events (participants affected / at risk) | 134/164 | 142/166 | 140/165 | 124/165 | 19/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK1437173A _LD Group (N=164) | GSK1437173A _MD Group (N=166) | GSK1437173A _HD Group (N=165) | Placebo + GSK1437173A _HD Group (N=165) | Placebo Group (N=54)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 2 (2) | 4 (4) | 3 (3) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia supraventricular (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradyarrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Cardiac failure (Cardiac disorders) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Right ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinoatrial block (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal angiodysplasia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retinal vein thrombosis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic gastropathy (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Intestinal polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peptic ulcer perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal prolapse (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cyst (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device dislocation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drowning (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Medical device complication (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Allergy to arthropod bite (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amyloidosis (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Clostridial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic gangrene (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Febrile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis aeromonas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis clostridial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lymphangitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuroborreliosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Pneumonia primary atypical (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis aspergillus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Asbestosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meniscus lesion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skull fractured base (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tooth injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bone cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 5 (5) | 3 (3) | 1 (1)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemangiopericytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypopharyngeal cancer stage iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Melanoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dementia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drop attacks (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Partial seizures (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (2) | 0 (0) | 2 (2) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Vascular encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viith nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Glomerulonephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oliguria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femoral arterial stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK1437173A _LD Group (N=164) | GSK1437173A _MD Group (N=166) | GSK1437173A _HD Group (N=165) | Placebo + GSK1437173A _HD Group (N=165) | Placebo Group (N=54)
Erythema (Skin and subcutaneous tissue disorders) | 68 (91) | 65 (102) | 68 (96) | 50 (50) | 2 (4)
Fatigue (General disorders) | 69 (92) | 85 (118) | 73 (99) | 47 (58) | 12 (17)
Headache (Nervous system disorders) | 48 (65) | 60 (73) | 51 (64) | 36 (40) | 9 (14)
Myalgia (Musculoskeletal and connective tissue disorders) | 75 (109) | 89 (128) | 70 (105) | 49 (57) | 9 (13)
Pain (General disorders) | 115 (193) | 121 (205) | 122 (199) | 93 (95) | 9 (11)
Pyrexia (General disorders) | 20 (21) | 19 (21) | 22 (23) | 9 (9) | 0 (0)
Swelling (General disorders) | 43 (55) | 32 (43) | 45 (54) | 30 (30) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.